CLINICAL TRIAL: NCT02129725
Title: Renin- Angiotensin and Fibrinolysis Interaction in Humans: Effect of Long-term PDE-5 Inhibition on Glucose Homeostasis. Sub-study
Brief Title: Effect of Prolonged PDE-5 Inhibition on Insulin Signaling in Skeletal Muscle.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, Professor Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 110206-substudy
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sildenafil citrate (Experimental): In the parent study, subjects are randomized to sildenafil 25 mg tid.
  Interventions: Drug: Sildenafil citrate
- placebo oral capsule (Placebo Comparator): In the parent study, subjects are randomized to matching placebo
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Sildenafil citrate — Sildenafil citrate 25 mg, 1 capsule three times a day for 3 months
  Other Names: Viagra
  Arms: sildenafil citrate
Drug: Placebo Oral Capsule — placebo capsules, 1 capsule po three times a day for 3 months
  Other Names: placebo comparator
  Arms: placebo oral capsule

SUMMARY:
Our research proposal will determine if PDE-5 inhibition exerts a favorable effect on insulin signaling pathways in skeletal muscle of subjects with impaired fasting glucose and/or impaired glucose tolerance.

DETAILED DESCRIPTION:
Participants enrolled in the study titled " Renin-angiotensin and fibrinolysis interaction in humans: effect of long-term PDE5 inhibition on glucose Homeostasis, (Specific aim 2)" will be offered the opportunity to participate in this sub-study.

We will obtain skeletal muscle biopsies from 16 subjects who are enrolled in specific aim 2. Eight subjects will be in the sildenafil group and 8 subjects will be in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years and BMI > 25 kg/M2 (> 23 kg/M2 among Asian Americans) and ≤40kg/m2 Impaired fasting glucose (100-125mg/dL) and/or impaired glucose tolerance (2-hr plasma glucose 140-199 mg/dL) and/or hemoglobin A1c 5.7-6.4%

Exclusion Criteria:

* Diabetes type 1 or type 2, as defined by a fasting glucose of 126 mg/dL or greater, a two-hour plasma glucose of 200 mg/dL or greater, or the use of anti-diabetic medication.
* The use of nitrates or any disease that might require the use of nitrates.
* The use of any potent CYP3A4 inhibitor.
* Subjects who have participated in a weight-reduction program during the last 6 month or whose weight has increased or decreased more than 2 kg over the preceding 6 months.
* Pregnancy. Women of child-bearing potential will be required to have undergone tubal ligation or to be using barrier or hormonal methods of birth control.
* Breast-feeding.
* Cardiovascular disease such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure, deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy.
* Treatment with anticoagulants.
* Treatment with metformin.
* History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack.
* History or presence of immunological or hematological disorders.
* Diagnosis of asthma on current inhaled corticosteroid therapy.
* Clinically significant gastrointestinal impairment that could interfere with drug absorption.
* Impaired hepatic function (aspartate amino transaminase and/or alanine amino transaminase >1.5 x upper limit of normal range)
* Impaired renal function (serum creatinine >1.5 mg/dl).
* Hematocrit <35%.
* Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult.
* Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month).
* Treatment with lithium salts.
* History of alcohol or drug abuse.
* Treatment with any investigational drug in the 1 month preceding the study.
* Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study.
* Inability to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects consented to give muscle biopsy
Groups:
- Sildenafil: In the parent study, subjects are randomized to sildenafil 25 mg tid.
  muscle biopsy: A muscle biopsy will be obtained before and after the hyperinsulinemic clamp in the parent study. The purpose of the biopsy will be to assess Akt signaling.
- Placebo: In the parent study, subjects are randomized to matching placebo
  muscle biopsy: A muscle biopsy will be obtained before and after the hyperinsulinemic clamp in the parent study. The purpose of the biopsy will be to assess Akt signaling.
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 8 | 7
Completed | 6 | 4
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: Subjects who consented (16) and were randomized (15).
Groups:
- Sildenafil; Placebo: Subjects consented for the biopsy substudy and randomized
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (12.8) | 47.3 (12.4) | 47.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15
Body mass index [Mean (Standard Deviation); unit: mg/kg2] | 31.5 (4.1) | 34.5 (5.0) | 32.9 (4.7)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 97.2 (10.3) | 91.4 (13.4) | 94.5 (11.7)
Two-hour glucose [Mean (Standard Deviation); unit: mg/dL] | 122.6 (45.4) | 134.3 (37.9) | 128.0 (41.0)

OUTCOME MEASURES:

1. Primary Outcome: Insulin-stimulated AKT Phosphorylation
Description: measured using Western blot for pAkt and for total Akt from muscle biopsies obtained at the end of the baseline hyperinsulinemic clamp and the three-month hyperglycemic clamp.
  The ratio of pAkt to Akt expression was calculated at each time point and the change in ratio from 0 to 3 months is presented.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: change in ratio
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 6 | 4
change in ratio | 0.065 (0.160) | -0.457 (0.710)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Sildenafil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 5/8 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=8) | Placebo (N=7)
pain at biopsy site (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
bleeding at biopsy site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 0 (0)
low potassium (Renal and urinary disorders) | 1 (1) | 0 (0)
joint or muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — not at biopsy site
vasovagal episode (Cardiac disorders) | 0 (0) | 1 (1)
flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
palpitations (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes